CLINICAL TRIAL: NCT02643199
Title: Automated Fetal Heart Echocardiography by Five-Dimensional Ultrasound in the Third Trimester of Pregnancy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Lecturer of Obstetrics and Gynaecology Faculty of Medicine, Ain Shams University, Ain Shams University
Other Study IDs: 5D Echocardiography
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Fetal Heart Echocardiography by Five Dimensional Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study to evaluate Five-Dimensional Ultrasound in automated assessment of the fetal heart from 20-36 weeks of gestation.

DETAILED DESCRIPTION:
This is a Prospective pilot study that will be performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.

90 pregnant women will be recruited from the Fetal Care Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.

All cases will be subjected to:

1. Full history taking including patient's age, parity, last menstrual period, estimated gestational age by dates, past history of medical disorders, clinical examinations (General and abdominal).
2. Two-Dimensional Ultrasound and Five-Dimensional Ultrasound will be done for all cases for assessment of fetal Heart.

   * 90 consecutive patients will undergo 2D fetal echocardiography by one observer
   * Then they will undergo blindly Five-Dimensional fetal echocardiography by another observer
   * The data collected will be compared to evaluate the accuracy of Five-Dimensional US in fetal heart assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. Gestational age at 34-36 weeks as determined be date and last menstrual period.
3. Normal Amniotic Fluid Index.

Exclusion Criteria:

1. Multiple pregnancies.
2. Oligohydramnios or Polyhydramnios (AFI > 95th percentile or < 5th percentile).
3. Obese patient, BMI > 30
4. Intrauterine growth restriction.
5. Fetal spine between the 11- and 1- O'clock positions due to possibility of shadowing from ribs or spine

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a Prospective pilot study that will be performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.
  Ninety pregnant women will be recruited from the Fetal Care Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Automated Fetal Heart Echocardiography by Five-Dimensional Ultrasound in the Third Trimester of Pregnancy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Prospective pilot study that was performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.
  90 pregnant women were recruited from the Fetal Care Unit who will fulfill the inclusion criteria.
Groups:
- Pregnant Women From 20 to 36 Weeks of Pregnancy: This is a Prospective pilot study that was performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.
  90 pregnant women were recruited from the Fetal Care Unit who will fulfill the inclusion criteria.
  Two-Dimensional Ultrasound and Five-Dimensional Ultrasound were done for all cases for assessment of fetal Heart.
Period: Overall Study
Arm/Group | Pregnant Women From 20 to 36 Weeks of Pregnancy
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant Women From 20 to 36 Weeks of Pregnancy
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Satisfactory Fetal Echocardiography Views by Two-Dimensional Ultrasound
Description: Fetal Echocardiography by Two-Dimensional Ultrasound measurement was done to examine fetal heart in both sagittal Views and transverse views:
  1. Four chamber view
  2. Five chamber view
  3. Left outflow tract
  4. Right outflow tract
  5. 3 vessels and Trachea View
  6. Abdomen/Stomach
  7. Ductal arch
  8. aortic arch
  9. Bicaval view then we count howmuch views of nine views were satisfactory
Time Frame: 20 - 36 weeks of gestation
Measure: Mean (Standard Deviation); unit: Number of satisfactory views
Arm/Group | Pregnant Women From 20 to 36 Weeks of Pregnancy
Number analyzed (Participants) | 90
Number of satisfactory views | 8.7 (0.8)

2. Secondary Outcome: Number of Satisfactory Fetal Echocardiography Views by Five-Dimensional Ultrasound
Description: Fetal Echocardiography by Five-Dimensional Ultrasound measurement was done to examine fetal heart in both sagittal Views and transverse views:
  1. Four chamber view
  2. Five chamber view
  3. Left outflow tract
  4. Right outflow tract
  5. 3 vessels and Trachea View
  6. Abdomen/Stomach
  7. Ductal arch
  8. aortic arch
  9. Bicaval view then we count howmuch views of nine views were satisfactory
Time Frame: 20 - 36 weeks of gestation
Measure: Mean (Standard Deviation); unit: Number of satisfactory views
Arm/Group | Pregnant Women From 20 to 36 Weeks of Pregnancy
Number analyzed (Participants) | 90
Number of satisfactory views | 8.9 (0.4)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Two-Dimensional Ultrasound and Five-Dimensional Ultrasound were performed and adverse Events Adverse Events were assessed.
Arm/Group | Pregnant Women From 20 to 36 Weeks of Pregnancy
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No